CLINICAL TRIAL: NCT04722640
Title: Exploring the Effects of IL-23 Inhibition by Risankizumab on Psoriasis Autoimmunity
Acronym: PSORIASI_RISA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2763
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RISAKIZUMAB (Experimental): SKYRIZI
  Interventions: Drug: SKYRIZI

INTERVENTIONS:
Drug: SKYRIZI — SKYRIZI

SUMMARY:
Approximately 80 patients affected by moderate to severe psoriasis will be screened for the presence of LL37( and ADAMTSL5 autoreactive T-cells in their blood at Day 0. Patients whose lymphocytes reacted with proliferation to LL37 or ADAMTSL5 will receive SKYRIZI (Risakizumab) at Day 1, week 4, 16, 28, 40. LL37 and ADAMTSL5-specific T-cell responses will be evaluated at Day 0, week 16, week 28 and week 52. Each patient will be followed for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent
2. Subject is > 18 and < 75 years of age at time of screening
3. Subject has had stable moderate to severe plaque psoriasis for at least 6 months (e.g., no morphology changes or significant flares of disease activity in the opinion of the Investigator)
4. Subject has involved body surface area (BSA) > 10% and PASI > 12 at baseline
5. Subject candidates to SKYRIZI therapy according to local label
6. Subject is able to complete study procedures, including self-assessments and self injections
7. Subjects who responded with T-lymphocytes proliferation to the psoriasis autoantigen LL37 or ADAMTSL5.
8. Subject is male or a woman not of child-bearing potential, including:

   1. infertile patients due to surgical sterilization, congenital anomalies
   2. OR postmenopausal, defined as: a woman of at least 50 years of age with an intact uterus, not on hormone therapy, who has either:

      * Cessation of menses for at least 1 year
      * OR At least 6 months of spontaneous amenorrhea with a follicle stimulating hormone level of >40 mIU/mL
   3. OR A woman of 55 years or older not on hormone therapy who has had at least 6 months of spontaneous amenorrhea
   4. OR A woman at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy
9. Subject is a woman of child-bearing potential and:

   1. Must test negative for pregnancy prior to first dose in Study
   2. Must agree to either remain abstinent, if complete abstinence is their preferred and usual lifestyle, or remain in same-sex relationships, if part of their preferred and usual lifestyle, or without sexual relationships with males. Periodic abstinence (for example, calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence just for the duration of a trial, and withdrawal are not acceptable methods of contraception.
   3. OR Must use 2 effective methods of contraception for the entirety of the study. Abstinence or contraception must continue for 21 weeks following completion of investigational product administration

      * Two effective methods of contraception (such as male or female condoms with spermicide, diaphragms with spermicide or cervical sponges) will be used. The patient may choose to use a doublebarreled method of contraception. Barrier protection methods without concomitant use of a spermicide are not a reliable or acceptable method. Thus, each barrier method must include use of a spermicide. It should be noted that the use of male and female condoms as a double-barrier method is not considered acceptable due to the high failure rate when these methods are combined.
      * Of note, 1 of the 2 methods of contraception may be a highly effective (less than 1% failure rate) method of contraception (such as, combination oral contraceptives, implanted contraceptives or intrauterine devices).

Exclusion Criteria:

Skin disease related:

1. Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions at the time of the screening visit (e.g., eczema) that would interfere with evaluations of the effect of investigational product on psoriasis

   Other medical conditions:
2. Subject has a planned surgical intervention during the duration of the study
3. Subject has a known history of human immunodeficiency virus
4. Hepatitis B surface antigen or Hepatitis C antibody positivity at screening
5. Patient is hepatitis B core antibody positive (HBcAb+) but HbsAg and HBsAb negative
6. Subject has uncontrolled, clinically significant systemic disease such as diabetes mellitus, cardiovascular disease, renal failure, liver disease, or hypertension
7. Subject has any active malignancy, including evidence of cutaneous basal orsquamous cell carcinoma or melanoma
8. Subject has history of malignancy within 5 years except treated and considered cured cutaneous squamous or basal cell carcinoma, in situ cervical cancer, or in situ breast ductal carcinoma
9. Subject has any concurrent medical condition that, in the opinion of the Investigator, could cause this study to be detrimental to the subject
10. Has active TB or other serious infection
11. Has received, or is expected to receive, any live virus or bacterial vaccination within 4 weeks before the first administration of study intervention

    Laboratory abnormalities:
12. Laboratory abnormalities at screening, including any of the following:

    * Hemoglobin < 9 g/dL
    * Platelet count < 100,000/mm3
    * White blood cell count < 3,000 cells/mm3
    * Absolute neutrophil count (ANC) < 1000/mm3
    * Creatinine clearance < 50 mL/min (Cockcroft-Gault formula)
    * Any other laboratory abnormality, which, in the opinion of the Investigator, will prevent the subject from completing the study or will interfere with the interpretation of the study results

    Washouts and non-permitted drugs:
13. Has received prior treatment with IL-12/23 inhibitor or IL23 inhibitor. Has received any with other biological agents for psoriasis without proper washout period of 4 weeks.
14. Subject has used UV B therapy within 14 days before first dose of investigational product
15. Subject has used topical therapy for psoriasis as follows:

    * superpotent (class I) or potent (class II) topical steroids or topical anthralin within 14 days before first dose of investigational product
    * any other formulation or potency of topical therapy or UV B phototherapy within 14 days before first dose of investigational product (exception: upper mid-strength to least potent [class III to VII] topical steroids permitted on the palms, soles, face and intertriginous areas)
16. Subject has used the following within 28 days of first dose of investigational product:

    * UVA light therapy (with or without psoralen) or excimer laser;
    * non-biologic systemic therapy for psoriasis (including but not limited to oral retinoids, cyclosporine, systemically administered calcineurin inhibitors, azathioprine, thioguanine, hydroxyurea, fumarates, or oral or parenteral corticosteroids including intramuscular or intraarticular administration [exception: optic, nasal, or inhaled corticosteroids within recommended doses is permitted])
17. Subject currently is enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s) General
18. Active substance abuse (within 24 weeks of screening)
19. Has known intolerance or hypersensitivity to Risakizumab, or known allergies or clinically significant reactions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of activated autoantigen-specific T-cells | 12 Months
  Proportion of activated autoantigen-specific T-cells as measured by LL37 and ADAMTSL5 antigens by antigenic-specific proliferation assay at 28 weeks with respect to baseline.

IPD SHARING:
Plan to Share IPD: No